CLINICAL TRIAL: NCT04120649
Title: Comparison Between Different Risk Stratification Models for Prediction of Lymph Node Involvement in Endometrial Carcinoma
Brief Title: Different Risk Stratification Models for Prediction of Lymph Node Involvement in Endometrial Carcinoma
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: RSMLI
Record Dates: First submitted 2019-10-06; First posted 2019-10-09 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endomterial cancer: All patients visiting the clinic at Women Health Hospital who having endometrial carcinoma with their diagnosis based on investigations (tumor marker ) , imaging, histopathology will have surgical staging consisted of total hysterectomy, bilateral salpingo-oopherectomy (based on the age of the patient), pelvic and para-aortic lymphadenectomy, and peritoneal washings
  Interventions: Procedure: hysterectomy

INTERVENTIONS:
Procedure: hysterectomy — total hysterectomy, bilateral salpingo-oopherectomy (based on the age of the patient), pelvic and para-aortic lymphadenectomy, and peritoneal washings

SUMMARY:
Endometrial cancer is the most common malignant disease of the female genital tract and the seventh most common cause of cancer death in women in Western countries. Histological type, grade and depth of myometrial invasion are prognostic factors in early stage disease as well as risk factors for lymph node metastasis. Systematic lymphadenectomy has recently been questioned for stage I disease based on the results from two randomized trials

ELIGIBILITY:
Inclusion Criteria:

* Not virgin
* Not having congenital anomalies
* Early stage
* Body mass index less than 35

Exclusion Criteria:

* virgin
* advanced stage
* sever infection especially in the pelvis
* lymphadenopathy for any cause
* lymphadenectomy for any cause
* BMI more than 35
* Synchronous malignancies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who having endometrial carcinoma
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
the validity of Mayo criteria risk stratification model | 3 months
  risk stratification model for prediction of lymph node involvement in women with endometrial carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt